CLINICAL TRIAL: NCT02668406
Title: Establishment of a Reference Clinical Sample Panel Allowing for the Development and Proof-of-concept Validation of an In-vitro Diagnostic Test for the Diagnosis of Melioidosis
Brief Title: Study to Obtain Blood and Voided Urine Samples to Improve the Diagnosis of Melioidosis
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Sihanouk Hospital Center of HOPE (Other); SRI International (Industry)
Responsible Party: Sponsor
Other Study IDs: Melioidosis
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Melioidosis; Systemic Inflammatory Response Syndrome; Suspected or Confirmed Bloodstream Infections
Keywords: Blood infection, melioidosis, rapid diagnostic test
MeSH Terms: conditions — Melioidosis; Systemic Inflammatory Response Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (phase A and B) and voided urine samples (only phase A)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Burkholderia pseudomallei: Patients for whom blood cultures grew Burkholderia pseudomallei
  Interventions: Other: Venous blood sampling (2 timepoints) (Phase A and B); Other: Voided urine sampling (first sample) (Phase A); Other: Voided urine sampling (second sample) (Phase A)
- No pathogen: Patients for whom blood cultures did not grow a pathogen, but have other body site grown with Burkholderia pseudomallei, or are suspected of melioidosis
  Interventions: Other: Venous blood sampling (2 timepoints) (Phase A and B); Other: Voided urine sampling (first sample) (Phase A); Other: Voided urine sampling (second sample) (Phase A)
- Another pathogen: Patients for whom blood cultures grew another pathogen
  Interventions: Other: Venous blood sampling (1 timepoint) (Phase A and B); Other: Voided urine sampling (first sample) (Phase A)

INTERVENTIONS:
Other: Venous blood sampling (2 timepoints) (Phase A and B) — 8.5ml at Day 1 + 8.5ml at Day 5
  Groups: Burkholderia pseudomallei; No pathogen
Other: Venous blood sampling (1 timepoint) (Phase A and B) — 8.5ml at Day 1
  Groups: Another pathogen
Other: Voided urine sampling (first sample) (Phase A) — At least 20ml upon confirmation of being part of one of the 3 study groups
Other: Voided urine sampling (second sample) (Phase A) — At least 20ml during routine hospital stay or routine follow-up visit
  Groups: Burkholderia pseudomallei; No pathogen

SUMMARY:
Clinical samples [blood and voided urine (only for phase A)] from patient recruited at Sihanouk Hospital Centre of HOPE (SHCH) and HOPE Community Medical Center (CMC) will be processed (decontamination) and shipped to SRI International with the purpose of design and validation (proof of concept) and (case/control series) of in-vitro diagnostics for melioidosis.

DETAILED DESCRIPTION:
Study will be proposed to all patients at Sihanouk Hospital Centre of HOPE (SHCH) and HOPE Community Medical Center (CMC) presenting with systemic inflammatory response syndrome (SIRS).

Blood samples will be collected upon admission for patients with blood culture request as part of routine patient care and agreement on informed consent. A second sample will be collected in patients with blood culture proven melioidosis or suspicion of melioidosis (only for phase B), at day 5 after initiation of appropriate antibiotic treatment. Depending on the final diagnosis, a subset of patients will be assigned to 3 groups:

1. Patients for whom blood cultures grew Burkholderia pseudomallei
2. Patients for whom blood cultures did not grow a pathogen, but have other body site grown with Burkholderia pseudomallei, or are suspected of melioidosis
3. Patients for whom blood cultures grew with another pathogen

In phase A only, at least 20 ml of voided urine will be collected when a patient is hospitalized and identified as belonging to study group 1, 2 or 3. A second collection of voided urine will be collected for group 1 and 2 patients during routine further hospital stay or a routine follow-up visit.

The clinical samples from these patients will be processed and shipped to SRI International with the purpose of design (=phase A) and validation (=phase B) of in-vitro diagnostics for melioidosis.

A coded database will be completed with basic demographic, clinical and microbiological data and final diagnosis. This coded information will be provided to SRI International.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old)
* Blood culture request by treating physician as part of standard care
* Willing to give informed consent

Exclusion Criteria:

* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with systemic inflammatory response syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 4203 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical reference panel (blood) | 15 months
  Establishment of a quality-assured and well-documented clinical reference panel (cases/control) of human blood samples allowing for the design, development and proof-of-concept validation of an in-vitro diagnostic assay for the diagnosis of melioidosis.
Clinical reference panel (urine) | 15 months
  Establishment of a quality-assured and well-documented clinical reference panel (cases/control) of human voided urine samples allowing for the design, development and proof-of-concept validation of an in-vitro diagnostic assay for the diagnosis of melioidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jacobs, MD, Study Director — Institute of Tropical Medicine, Antwerp, Belgium; Thong Phe, MD, Principal Investigator — Sihanouk Hospital Center of HOPE (SHCH), Cambodia
Locations (2):
- Cambodia (2):
  - HOPE Community Medical Center, Phnom Penh
  - Sihanouk Hospital Center of HOPE (SHCH), Cambodia, Phnom Penh